CLINICAL TRIAL: NCT06397157
Title: Combined Effects of Virtual Reality and Motor Imagery With Routine Physical Therapy in Patients With Non-specific Neck Pain
Brief Title: Combined Effects of Virtual Reality and Motor Imagery in Patients With Non-specific Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/02104
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cervical Pain; Kinesiophobia; Pain
Keywords: Cervical pain; Kinesiophobia; Pain; Motor Imagery; Virtual Reality
MeSH Terms: conditions — Neck Pain; Kinesiophobia; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality+Motor Imagery+Routine physical therapy (Experimental): Participants in Group A will receive Virtual Reality (VR) and Motor Imagery (MI) training with Routine physical therapy for every alternate day (3 days per week) for 6 weeks. Total number of sessions will be 18.
  Interventions: Other: Virtual Reality; Other: Motor Imagery; Other: Routine Physical therapy
- Virtual Reality+Routine physical therapy (Active Comparator): Participants in Group A will receive Virtual Reality (VR) training with Routine physical therapy for every alternate day (3 days per week) for 6 weeks. Total number of sessions will be 18.
  Interventions: Other: Virtual Reality; Other: Routine Physical therapy
- Motor Imagery+ Routine physical therapy (Active Comparator): Participants in Group A will receive Motor Imagery(MR) training with Routine physical therapy for every alternate day (3 days per week) for 6 weeks. Total number of sessions will be 18.
  Interventions: Other: Motor Imagery; Other: Routine Physical therapy

INTERVENTIONS:
Other: Virtual Reality — Participants will recieve treatment(Virtual reality) for every alternate day (3 days per week) for 6 weeks. Total number of sessions will be 18.
  Arms: Virtual Reality+Motor Imagery+Routine physical therapy; Virtual Reality+Routine physical therapy
Other: Motor Imagery — Participants will recieve treatment(Motor Imagery) for every alternate day (3 days per week) for 6 weeks. Total number of sessions will be 18.
  Arms: Motor Imagery+ Routine physical therapy; Virtual Reality+Motor Imagery+Routine physical therapy
Other: Routine Physical therapy — Participants will recieve treatment(Routine physical therapy) for every alternate day (3 days per week) for 6 weeks. Total number of sessions will be 18.

SUMMARY:
Non-specific neck pain is the most common musculoskeletal symptom which can cause limited cervical mobility, impaired functional status and stress at work. Virtual reality and motor imagery are unique technologies which have beneficial effects on the treatment of non-specific neck pain. Virtual reality is a simulated 3D environment that enables users to explore and interact with a virtual surrounding while motor imagery (MI) is a dynamic mental process of an action, without its actual motor execution. This study aims to investigate the combined effects of Virtual Reality (VR) and Motor Imagery Techniques (MI) with Routine Physical Therapy (RPT) in patients with Non-specific neck pain. This randomized clinical trial will be carried at Railway General Hospital, Rawalpindi on 93 participants meeting the inclusion criteria included in the study through probability convenience sampling technique. 3 groups of participants assigned ramdomly will receive interventions for three days a week for 6 weeks. Group A will receive virtual reality (VR) and motor imagery (MI) along with routine physical therapy for . Group B participants will receive VR along with routine physical therapy while Group C will receive MI along with routine physical therapy. Total treatment time will be 40 minutes. Outcome measure tools will be Numeric pain rating scale to measure pain, the Tampa scale of Kinesiophobia (TSK) for the measurement of kinesiophobia and Neck disability index for disability and functional status.

DETAILED DESCRIPTION:
Non-specific neck pain is the most common musculoskeletal symptom which can cause limited cervical mobility, impaired functional status and stress at work. Despite of the duration, neck pain can impair functional capacity, quality of life and can cause worry, anxiety and depression. Virtual reality and motor imagery are unique technologies which have beneficial effects on the treatment of non-specific neck pain. Virtual reality is a simulated 3D environment that enables users to explore and interact with a virtual surrounding while motor imagery (MI) is a dynamic mental process of an action, without its actual motor execution. This study aims to investigate the combined effects of Virtual Reality(VR) and Motor Imagery Techniques (MI) with Routine Physical Therapy (RPT) in patients with Non-specific neck pain.

This randomized clinical trial will be carried at Railway General Hospital ,Rawalpinidi .93 participants meeting the inclusion criteria will be included in this study through a non-probability convenience sampling technique.

Participants will be randomly assigned into 3 groups using computer generated method. All the groups receive interventions for three days a week for 6 weeks. Group A will receive virtual reality (VR) and motor imagery (MI) along with routine physical therapy for . Group B participants will receive VR along with routine physical therapy while Group C will receive MI along with routine physical therapy. Total treatment time will be 40 minutes.

Outcome measure tools will be Numeric pain rating scale to measure pain, the Tampa scale of kinesiophobia (TSK) for the measurement of kinesiophobia and Neck disability index for disability and functional status. The data will be collected at baseline before the treatment of the patient, Follow-up on the 3rd week and post treatment measure on the 6th week to measure the outcome measures. Data will be analysed by SPSS version 26. Statistical significance will be set at p=0.05. The normality of data will be checked by using Kolmogorov- Smirnov test. For the between group analysis of parametric data, one way ANOVA will be used, while Kruskal-Wallis test will be applied for non-parametric data. For within group comparison repeated measure ANOVA will be applied for parametric data, for non-parametric data Friedman ANOVA will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patients should be 18-50 years
* Both females and males are included
* Patient should have a consistent pain for 3 months or more.
* Patient having non-specific neck pain.

Exclusion Criteria:

* Specific neck pain caused by metastasis, neoplasia, infectious or inflammatory disorders, bone fractures or traumatic precedents with neck injuries (2)
* Positive neurological signs or evidence of spinal compression (abnormal diffuse sensitivity, hyperreflexia, or diffuse weakness)
* Cervical osteoarthritis
* Spondylarthritis
* Neck pain associated with vertigo (vestibular involvement)
* Neck pain associated with whiplash injuries
* Previous cervical surgeries (2)
* Headaches before the onset of neck pain and without cervical origin
* Inability to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 6 weeks
  In a Numerical Pain Rating Scale (NRS), patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Zero usually represents no pain at all whereas the upper limit represents 'the worst pain ever possible'. Numerical Pain Rating Scales have shown high correlations with other pain-assessment tools in several studies.
The Tampa Scale for Kinesiophobia (TSK) | 6 weeks
  The Tampa Scale for Kinesiophobia (TSK) is a 17-item questionnaire that quantifies fear of movement. The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible Kinesiophobia, and the higher scores indicate an increasing degree of Kinesiophobia.
Neck Disability Index (NDI) | 6 weeks
  A modification of the Oswestry Low Back Pain Index was conducted producing a 10-item scaled questionnaire entitled the Neck Disability Index (NDI) for the measurement of disability and functional status. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. All section scores are then totaled. Scoring is reported on a 0-50 scale, 0 being the best possible score and 50 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M phil, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital ,Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kragting M, Voogt L, Coppieters MW, Pool-Goudzwaard AL. Visual feedback manipulation in virtual reality to influence pain-free range of motion. Are people with non-specific neck pain who are fearful of movement more susceptible? PLoS One. 2023 Jul 5;18(7):e0287907. doi: 10.1371/journal.pone.0287907. eCollection 2023. PMID 37406021
- [Background] Tejera DM, Beltran-Alacreu H, Cano-de-la-Cuerda R, Leon Hernandez JV, Martin-Pintado-Zugasti A, Calvo-Lobo C, Gil-Martinez A, Fernandez-Carnero J. Effects of Virtual Reality versus Exercise on Pain, Functional, Somatosensory and Psychosocial Outcomes in Patients with Non-specific Chronic Neck Pain: A Randomized Clinical Trial. Int J Environ Res Public Health. 2020 Aug 16;17(16):5950. doi: 10.3390/ijerph17165950. PMID 32824394
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Kortlever JTP, Tripathi S, Ring D, McDonald J, Smoot B, Laverty D. Tampa Scale for Kinesiophobia Short Form and Lower Extremity Specific Limitations. Arch Bone Jt Surg. 2020 Sep;8(5):581-588. doi: 10.22038/abjs.2020.40004.2073. PMID 33088859
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034